CLINICAL TRIAL: NCT01135160
Title: Evaluation of Weight Bearing in Patients After Total Hip and Knee Replacement
Brief Title: Evaluation of Weight Bearing After Total Hip and Knee Replacement
Status: Terminated | Type: Observational
Why Stopped: The planned number of patients was achieved.
Sponsor: Kantonsspital Münsterlingen (Other)
Responsible Party: Sponsor
Other Study IDs: KSM 2010-1
Record Dates: First submitted 2010-03-16; First posted 2010-06-02 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Arthropathy of Hip; Arthropathy of Knee
Keywords: weight bearing; pain; total hip arthroplasty; total knee arthroplasty; weight bearing after TKA or THA
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TKA/THA: All patients receiving TKA/THA meeting inclusion but not exclusion criteria

SUMMARY:
The regime in the aftercare after total hip and knee arthroplasty(THA/TKA) differs a lot between orthopedic surgeons concerning weight bearing. The type of implant and the way of implants' anchoring are considered.

In the literature there is no data so far about the way patient take care of the recommended weight bearing during the first 6 weeks after THA and TKA.

Over a one year period starting August 2010 all patients undergoing TKA or THA at the investigators institution will have a technical device in their shoes (sole) to measure the load in each step they do in these shoes during the first 6 weeks. Patients are asked to fill out a standardised pain protocol every day (VAS) and document need of pain medication. The investigators recommend 20kg of weight on the operated leg for 6 weeks and full weight bearing at the end of week six.

The investigators believe that patients will adjust weight bearing to their level of pain and not to their surgeons recommendations.

ELIGIBILITY:
Inclusion Criteria:

* received a THA or TKA in the mentioned period of time
* is able to walk on crutches
* is able to understand our recommendations
* signed informed consent

Exclusion Criteria:

* not able to walk on crutches
* not able to understand our recommendations
* other deformities of lower limbs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients receiving TKA or THA at our institution between August 2010 and August 2011
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
full weight bearing allowed and accomplished end of 6th week | 6 weeks
  full weight bearing allowed and accomplished, documented by special soles with an electronic device, which will record weight bearing continuously on an USB stick

SECONDARY OUTCOMES:
pain under partial weight bearing (recommended) | 6 weeks
  Patients will have a official standardised pain diary and should document their pain and need of analgetics according to instructions given (VAS, "Schweizer Krebsliga") at least on a daily basis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schueler, Dr. med., Principal Investigator — Chief of the department for orthopedic surgery Kantonsspital Münsterlingen, Schweiz
Locations (1):
- Kantonsspital Münsterlingen, Münsterlingen, Thurgau, Switzerland